CLINICAL TRIAL: NCT06838429
Title: Effect of PARP Inhibitors Maintenance Therapy on the Survival Rate of Advanced or Relapsed Epitherlial Ovarian Cancer: an Observational Cohort Study
Brief Title: PARPi and Ovarian Cancer Survival
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Institute for Ovarian Cancer, Fudan University; Department of Gynecologic Oncology, Cancer Center, Fudan University Zhongshan Hospital, Shanghai, China (Unknown); Department of Gynecologic Oncology, Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, China (Unknown); Department of Gynecologic Oncology, State Key Laboratory of Oncology in South China, Collaborative Innovation Centre for Cancer Medicine, Sun Yat-sen University (Unknown); Department of Gynecologic Oncology, Fudan University Cancer Hospital, Shanghai, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: PARPi_OC
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Epithelial Ovarian Cancer, Fallopian Tube or Peritoneum; PARP Inhibitor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with newly diagnosed advanced epithelial ovarian cancer: Patients who were newly diagnosed with stage IIIC or IV primary epithelial ovarian cancer between December 2013 and December 2024.
- Patients with platinum-sensitive first relapsed epithelial ovarian cancer: Patients with platinum-sensitive first relapsed ovarian cancer who were diagnosed between December 2013 and December 2024

SUMMARY:
With the widespread use of PARP inhibitors (PARPi) as maintenance therapy in ovarian cancer, there is still a lack of real-world data from large samples regarding their impact on survival outcomes in advanced and recurrent ovarian cancer. This study aims to conduct a pragmatic cohort study to evaluate the impact of first-line and second-line maintenance treatment with PARPi on survival rates in patients with advanced and recurrent ovarian cancer. The genetic status, different PARPi drugs, and the use of anti-angiogenic inhibitor maintenance therapy or not is used as confounding factors.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Patients newly diagnosed with stage IIIC or IV primary epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer between December 2013 and December 2024.
* Complete data on first-line treatment and maintenance therapy.
* Availability of follow-up data.

Group 2:

* Patients with platinum-sensitive first recurrence of any stage of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, diagnosed between December 2013 and December 2024.
* Disease progression occurring at least 6 months after the completion of the last platinum-based chemotherapy regimen.
* Complete data on second-line treatment and maintenance therapy.
* Availability of follow-up data.

Exclusion Criteria:

Group 1:

* Non-epithelial tumors, borderline tumors, clear cell carcinoma, mucinous carcinoma.
* Missing first-line or follow-up data.

Group 2:

* Non-epithelial tumors, borderline tumors, clear cell carcinoma, mucinous carcinoma.
* Patients with second relapse.
* Platinum-resistant patients, such as those who had disease progression during chemotherapy or within 6 months after platinum-based chemotherapy.
* Missing second-line or follow-up data.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were newly diagnosed with stage IIIC or IV primary epithelial ovarian cancer or had platinum-sensitive first relapsed ovarian cancer between December 2013 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overall Mortality | 11 years
  Mortality of any cause